CLINICAL TRIAL: NCT05341258
Title: Arterial and End-Tidal CO2 Gradient as a Mortality Predictor in Critical Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3751
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-11

CONDITIONS: Critical Illness; Ventilation Perfusion Mismatch; Shock; Pulmonary Embolism; Trauma; Copd
MeSH Terms: conditions — Critical Illness; Shock; Pulmonary Embolism; Wounds and Injuries; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Critical Care Patients whom intubated last 24 hours (Other): Critical Care Patients whom intubated last 24 hours
  Interventions: Diagnostic Test: EtCO2; Diagnostic Test: PaCO2

INTERVENTIONS:
Diagnostic Test: EtCO2 — EtCO2
Diagnostic Test: PaCO2 — PaCO2

SUMMARY:
Scoring systems (SOFA, APACHE-II etc.) are used to estimate the mortality rates of patients treated in the intensive care unit. . In the scoring systems used, the disfunction level of the organs of the patients is measured. Blood gas analysis is routinely performed in patients whom intubated in the intensive care unit and receiving mechanical ventilation support, and the patient's treatment is optimized according to the results of the examination. The patient's mechanical ventilation settings are regulated by analyzing the Partial Arterial Carbondioxide (paCO2) value in the patient's blood gas result. The difference between the paCO2 value in the blood gas and the End-tidal Carbondioxide (EtCO2) value measured in the mechanical ventilator is 3-5mmHg in normal healthy people, while this difference is seen more in critical care patients. In critically ill patients in the intensive care unit, there is a greater increase in the difference between paCO2 and ETCO2 in cases where mortality is high, such as global perfusion disorder, shock situations, and massive pulmonary embolism, etc. In this study, it was planned to investigate the use of the difference between the paCO2 value in the blood gas taken from the patient and the ETCO2 value measured in the mechanical ventilator to predict the mortality rate of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Critical Care Patients intubated in last 24 hours.

Exclusion Criteria:

* Patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months
  Evaluation of correlation between PaCO2 and ETCO2 gradient difference and mortality in intubated critical care patients and mortality rates

SECONDARY OUTCOMES:
ICU Length of Stay | 6 months
  Days patients treated at ICU
Ventilator Free Days | 6 months
  Days during which the patient was mechanically ventilated

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Aygen Turkmen, Proffessor, Study Director — Director of Anesthesiology and Reanimation Department
Locations (1):
- Gaziosmanpasa Training Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No